CLINICAL TRIAL: NCT00092586
Title: A Multi-center, Double-Blind, Randomized, Placebo-Controlled, Parallel Group, 6-Week Study to Evaluate the Efficacy and Safety of Ezetimibe 10 mg/Day When Added to Ongoing Therapy With a Statin Versus Statin Therapy Alone, in Patients With Hypercholesterolemia Who Have Not Reached National Cholesterol Education Program (NCEP) Adult Treatment Panel (ATP) III Target LDL-Cholesterol Level
Brief Title: Study of an Approved Drug With a Statin (a Medication That Lowers Cholesterol Levels) as Compared to Statin Therapy Alone in Patients With High Cholesterol (0653-040)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653-040; 2004_037
Record Dates: First submitted 2004-09-23; First posted 2004-09-28 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0653, ezetimibe
Drug: Comparator: statins

SUMMARY:
The purpose of this 6-week study is to compare the reduction in specific levels of cholesterol in patients with high cholesterol.

DETAILED DESCRIPTION:
The duration of treatment is 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* High cholesterol levels that are identified by specific laboratory values

Exclusion Criteria:

* Active liver disease
* Any condition or situation which would interfere with participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2904 (Actual)
Dates: Start 2002-09; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Percent change in LDL-C

SECONDARY OUTCOMES:
Percentage of patients reaching NCEP ATP III target LDL-C levels

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Pearson TA, Denke MA, McBride PE, Battisti WP, Brady WE, Palmisano J. A community-based, randomized trial of ezetimibe added to statin therapy to attain NCEP ATP III goals for LDL cholesterol in hypercholesterolemic patients: the ezetimibe add-on to statin for effectiveness (EASE) trial. Mayo Clin Proc. 2005 May;80(5):587-95. doi: 10.4065/80.5.587. PMID 15887425
- [Background] Pearson T, Denke M, McBride P, Battisti WP, Brady WE, Palmisano J. Effectiveness of the addition of ezetimibe to ongoing statin therapy in modifying lipid profiles and attaining low-density lipoprotein cholesterol goals in older and elderly patients: subanalyses of data from a randomized, double-blind, placebo-controlled trial. Am J Geriatr Pharmacother. 2005 Dec;3(4):218-28. PMID 16503317
- [Background] Pearson TA, Denke MA, McBride PE, Battisti WP, Gazzara RA, Brady WE, Palmisano J. Effectiveness of ezetimibe added to ongoing statin therapy in modifying lipid profiles and low-density lipoprotein cholesterol goal attainment in patients of different races and ethnicities: a substudy of the Ezetimibe add-on to statin for effectiveness trial. Mayo Clin Proc. 2006 Sep;81(9):1177-85. doi: 10.4065/81.9.1177. PMID 16970214
- [Background] Denke M, Pearson T, McBride P, Gazzara RA, Brady WE, Tershakovec AM. Ezetimibe added to ongoing statin therapy improves LDL-C goal attainment and lipid profile in patients with diabetes or metabolic syndrome. Diab Vasc Dis Res. 2006 Sep;3(2):93-102. doi: 10.3132/dvdr.2006.020. PMID 17058629
- [Background] Pearson TA, Ballantyne CM, Veltri E, Shah A, Bird S, Lin J, Rosenberg E, Tershakovec AM. Pooled analyses of effects on C-reactive protein and low density lipoprotein cholesterol in placebo-controlled trials of ezetimibe monotherapy or ezetimibe added to baseline statin therapy. Am J Cardiol. 2009 Feb 1;103(3):369-74. doi: 10.1016/j.amjcard.2008.09.090. Epub 2008 Oct 30. PMID 19166691
- [Derived] Thongtang N, Lin J, Schaefer EJ, Lowe RS, Tomassini JE, Shah AK, Tershakovec AM. Effects of ezetimibe added to statin therapy on markers of cholesterol absorption and synthesis and LDL-C lowering in hyperlipidemic patients. Atherosclerosis. 2012 Dec;225(2):388-96. doi: 10.1016/j.atherosclerosis.2012.09.001. Epub 2012 Sep 13. PMID 23040830